CLINICAL TRIAL: NCT00894309
Title: Evaluation of the Validity of a New Index Provided by the PiCCO2 Device for Predicting Fluid Responsiveness in Critically Ill Patients
Brief Title: Validation of the Fluid Responsiveness Index in Critically Ill Patients
Acronym: FRI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bicetre Hospital (Other)
Responsible Party: Prof Jean-Louis TEBOUL, Medical Intensive Care Unit - Bicêtre Hospital
Other Study IDs: FRI-1
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-05

CONDITIONS: Shock; Critically Ill
MeSH Terms: conditions — Shock; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Fluid therapy is an important part of the management of patients with hemodynamic instability in the intensive care unit. By increasing cardiac preload, it aims at elevating cardiac output (CO) and thus restoring hemodynamic conditions in patients who are preload responsive. By contrast, volume administration can be deleterious in terms of pulmonary edema formation or other manifestations or fluid overload, especially in patients who are not preload responsive. Functional dynamic parameters that use heart-lung interactions, such as pulse pressure variation (PPV) and stroke volume variation (SVV) are considered accurate predictors of preload responsiveness in patients receiving fully controlled mechanical ventilation.

However, in cases of spontaneous breathing activity where heart-lung interaction indices fail to predict fluid responsiveness, one needs parameters able to reliably predict the hemodynamic response of fluid administration.

A new index that could indicate fluid responsiveness, so-called the fluid responsiveness index (FRI), has been elaborated. The advantage is that it could be used in patients who are not in control mechanical ventilation as well as in patients who are fully adapted to mechanical ventilation.

The FRI is based upon the analysis of continuous arterial and continuous central venous pressure. The FRI is determined by the relation of cardiac and respiratory activity; both are evaluated by means of power spectrum analysis of the pressures recorded.

The aim of this study is to test the value of the FRI to predict the hemodynamic response to fluid infusion in patients with hemodynamic instability not receiving fully controlled mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalization in an intensive care unit
* Presence of an acute circulatory failure as defined by the presence of at least one clinical sign of inadequate global perfusion
* Decision by the attending physician to give fluids will not be taken upon criteria predefined by the study protocol but considers:

  * systolic arterial pressure < 90 mmHg (or fall of systolic arterial pressure of more than 50 mmHg in known hypertensive patients)
  * urinary flow < 0.5 ml/kg/hr than two hours
  * tachycardia ≥ 100 beats/min
  * delayed capillary refill
  * mottled skin
  * high lactate
  * CO (Cardiac Output) that is not considered adequate and
  * low GEDV (Global EndDiastolic Volume)
* Monitoring by a PiCCO2™ device (Pulsion Medical Systems, Munich, Germany) already in place as part of the routine hemodynamic monitoring

Exclusion Criteria:

* Clinical evidence of pulmonary edema, hypervolemia or ELWI > 10 ml/kg

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an acute circulatory failure
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-05

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Monnet, MD, PhD, Principal Investigator — Medical Intensive Care Unit - Bicêtre Hospital; Azriel Perel, MD, PhD, Principal Investigator — Department of Anesthesiology and Intensive Care Sheba Medical Centre Tel Aviv; Jean-Louis Teboul, MD, PhD, Principal Investigator — Medical Intensive Care Unit - Bicêtre Hospital; Daniel Reuter, MD, PhD, Principal Investigator — Universitätsklinik Eppendorf, Hamburg; Wolfgang Huber, MD, PhD, Principal Investigator — II. Med. Klinik, Station 2/11, Munich; Fernando Suarez Sipmann, MD, PhD, Principal Investigator — Unidad de cuidados intensivos, Fundacion Jimenez Diaz, Madrid
Locations (5):
- Medical Intensive Care Unit, Le Kremlin-Bicêtre, France
- Germany (2):
  - Universitätsklinik Eppendorf, Hamburg
  - Klinikum Rechts der Isar, Munich
- Department of Anesthesiology and Intensive Care Sheba Medical Centre, Tel Aviv, Israel
- Unidad de cuidados intensivos, Fundacion Jimenez Diaz, Madrid, Spain